CLINICAL TRIAL: NCT04207866
Title: Evaluation of Teleconferencing in the Provision of Auditory Training Services
Brief Title: Auditory Training Via Teleconference
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Kassandra Kaminskas, Clinical Audiologist - Cochlear Implant Program, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 348-2019
Record Dates: First submitted 2019-10-25; First posted 2019-12-23 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Hearing Impairment, Sensorineural; Auditory; Nerve; Cochlear Implants; Rehabilitation
Keywords: Auditory Training; Teleconferencing
MeSH Terms: conditions — Hearing Loss, Sensorineural; Vestibulocochlear Nerve Diseases

STUDY DESIGN:
Intervention Model Description: The study is a prospective observational study with sequential enrolment of 40 cochlear implant recipients. The subjects will be continuously included in the study, and will be included in the teleconferencing or on-site groups based on willingness to travel and distance from the hospital. Individuals will first be assessed by an Audiologist to determine listening goals and provide structure for auditory training sessions in house. Follow-up sessions will involve TC or FTF sessions whereby the patient will work with a CDA on skills targeted to help the patient achieve listening goals. A review session may also occur with the Audiologist following several TC or FTF sessions to assess progress and reassess current goals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote AT services (Experimental): Experimental group will consist of participants who access auditory therapy services from a remote location. Services will be conducted with this group via teleconferencing over the Ontario Health Network.
  Interventions: Other: Teleconferencing; Other: Auditory training services
- In House AT (Active Comparator): This group will receive auditory therapy services face-to-face at the treatment site.
  Interventions: Other: Auditory training services

INTERVENTIONS:
Other: Teleconferencing — Use of video/audio stream to provide auditory training at a remote site.
  Arms: Remote AT services
Other: Auditory training services — Participants will engage in regular visits with a specialist to: 1) facilitate auditory training exercises; 2) work with the family/friends to encourage optimal communication strategies in the home; 3) evaluate and assess achievement of listening goals.
  Auditory training assess/reviews skills associated with but not necessarily limited to: 1) developing strategies to repair communication breakdowns; 2) listening in quiet; 3) listening in noise; 4) listening to a degraded signal.

SUMMARY:
Multi-channel cochlear implants have been highly successful in restoring speech understanding to individuals with severe-to-profound hearing loss. Optimal programs facilitate access to sound but do not necessarily result in optimal performance. Practiced listening with auditory inputs is required to retrain the brain to hear using a cochlear implant. In some cases exposure to sound in everyday listening is sufficient; however, in others there is a need for the provision of auditory training (AT) by a trained professional. In these cases it is important to have regular visits with a specialist to: 1) facilitate auditory training exercises; 2) work with the family/friends to encourage optimal communication strategies in the home; 3) evaluate and assess achievement of listening goals.

This study seeks to evaluate the feasibility of providing auditory training services remotely for patient populations located outside of Toronto. This study also seeks to evaluate interindividual perspectives regarding access and benefits of these services across remote and in person sessions.

DETAILED DESCRIPTION:
Individuals with severe-to-profound hearing impairment, who no longer benefit from hearing aids, are candidates for cochlear implantation. In many cases these devices provide access to sound and are successful in restoring speech understanding; however, there are instances where individuals might need additional assistance in the form of auditory training (AT). This study will involve comparison of two groups of individuals. Participants will be randomly assigned to the standard of care group OR the remote care group. Individuals who meet eligibility criteria will be contacted to assess their willingness to participate in additional auditory training (AT) sessions. These sessions will be conducted either face-to-face or via the Ontario Telehealth network as per random assignment. AT sessions will occur over the first 3 months following activation of the cochlear implant. Outcomes will be assessed using performance measures and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Newly implanted subjects who might need additional auditory training supports (e.g. long-term deafened, limited communication partners etc.)
* Post-lingual onset of hearing loss
* No cognitive deficits
* English must be their native language
* Willingness to use teleconferencing methods to obtain AT services and residing >1 hr away by car from the hospital
* Willingness to attend these appointments with a communication partner wherever possible

Exclusion Criteria:

* Onset of hearing loss prior to two years of age (prelingual hearing loss)
* Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array, as confirmed by medical examination and imaging including MRI
* Hearing loss of retro-cochlear or central origin
* Additional handicaps that would prevent participation in evaluations
* Unrealistic expectations on the part of the subject, regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure(s) and prosthetic device
* Active middle ear infection
* Unwillingness or inability of the candidate to comply with all investigational requirements
* History of radiation
* Patient concerns regarding their own technological skills and ability to use teleconferencing methods

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Teleconferencing for AT Services: In house questionnaire | 2 years
  In house questionnaire assessing benefits of using remote network for provision of services. Questionnaires asks several questions related to quality of audio-visual signal, ease of use, duration of appointments and whether or not the participants outcomes were achieved. Responses are on a likert scale (Strongly agree (1), agree, neutral, disagree, strongly disagree (5)). Higher scores mean a poorer outcome.

SECONDARY OUTCOMES:
Speech performance | 2 years
  A battery of tests is used within the standard of care provided to cochlear implant recipients. These tests are used as a gauge of performance with the device in the real world. The first test is the Arizona Biologic (AzBio) test which is assessed in quiet and at +5 dB SNR. It is scores in percentage of words correct. Higher scores are correlated with better outcomes.
Speech performance | 2 years
  A battery of tests is used within the standard of care provided to cochlear implant recipients. These tests are used as a gauge of performance with the device in the real world. The second test is the Hearing in Noise (HINT) test which is assessed in quiet and at +5 dB SNR. It is scores in percentage of words correct. Higher scores are correlated with better outcomes.
Speech performance | 2 years
  A battery of tests is used within the standard of care provided to cochlear implant recipients. These tests are used as a gauge of performance with the device in the real world. The third test is the Consonant-Nucleus-Consonant (CNC) word test which is assessed in quiet and at +5 dB SNR. It is scores in percentage of words correct. Higher scores are correlated with better outcomes.
Connection reliability of telepractice services | 2 years
  Given that the remote connection can be impacted by power supply etc. a count of signal interference/breakdowns will be made over the course of the study. Different mediums may be used to provide services (e.g. Ontario Telehealth Network, Zoom, Webx) in order to provide support to CI users in a convenient manner for them.
Subjective Perspectives on Auditory Training Benefits | 2 years
  Participants will complete an in-house questionnaire addressing perceived benefits of the services they received as well as an assessment of audiovisual quality, disturbances in the appointment etc. for the teleconferencing group. The questionnaire uses a likert scale using descriptors of agreement (i.e. Strongly agree (1), agree, neutral, disagree, strongly disagree (5)). A higher score indicates poorer outcomes.
Client Oriented Scale of Improvement (COSI) | 2 years
  The COSI is a well recognized subjective questionnaire used to assess pre/post-treatment improvement in listening. It will be used to assess the participants perceived benefit of treatment prior to their first Auditory training appointment and again once they are done receiving these services. It asks the listener to generate up to 5 listening goals. It then uses subjective assessment to assess their improvement as a % of change. Reporting is also completed using a likert scale with descriptors (Worse, No difference, slightly better, better, much better). Higher percentage and greater degree of change are associated with better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Kassandra H Kaminskas, M.Cl.Sc., Principal Investigator — Sunnybrook Health Sciences Centre - Clinical Audiologist
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bush ML, Thompson R, Irungu C, Ayugi J. The Role of Telemedicine in Auditory Rehabilitation: A Systematic Review. Otol Neurotol. 2016 Dec;37(10):1466-1474. doi: 10.1097/MAO.0000000000001236. PMID 27755363
- [Background] Cullington H, Kitterick P, DeBold L, Weal M, Clarke N, Newberry E, Aubert L. Have Cochlear Implant, Won't Have to Travel: Introducing Telemedicine to People Using Cochlear Implants. Am J Audiol. 2016 Oct 1;25(3S):299-302. doi: 10.1044/2016_AJA-16-0018. PMID 27768192